CLINICAL TRIAL: NCT03174977
Title: Pharmacokinetics Distribution of Raltegravir Using Radiolabeling in HIV-infected Patients by PET/MR: a Pilot Study.
Brief Title: Pharmacokinetics Distribution of Raltegravir by PET/MR
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-17586
Record Dates: First submitted 2017-03-03; First posted 2017-06-05 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-Raltegravir (Experimental)
  Interventions: Drug: 18F-Raltegravir

INTERVENTIONS:
Drug: 18F-Raltegravir — A single microdose of 18F-Raltegravir will be given to individuals currently being treated for HIV-1 with antiretroviral therapy.

SUMMARY:
This is a single-center drug distribution and pharmacokinetic study of a single microdose of 18F-raltegravir given to 10 HIV-infected subjects who are either taking or not taking a raltegravir-containing ART regimen. After administration of IV 18F-raltegravir, subjects will undergo PET/MRI in order to determine the distribution of radiolabeled drug through the lymphoreticular system and other tissues throughout the entire body.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* HIV infection
* Initiated a combination ART (HAART) regimen

Exclusion Criteria:

* Screening absolute neutrophil count <1,000 cells/mm3, platelet count <70,000 cells/mm3, hemoglobin < 8 mg/dL, estimated creatinine clearance <40 mL/minute, aspartate aminotransferase >100 units/L, alanine aminotransferase >100 units/L.
* Serious illness requiring hospitalization or parental antibiotics within the preceding 3 months.
* Any vaccination 2 weeks prior to baseline (Day 0) visit and throughout the study period.
* Concurrent treatment with immunomodulatory drugs, or exposure to any immunomodulatory drug in the preceding 16 weeks (e.g. corticosteroid therapy equal to or exceeding a dose of 15 mg/day of prednisone for more than 10 days, IL-2, interferon-alpha, methotrexate, cancer chemotherapy). NOTE: Use of inhaled or nasal steroid use is not exclusionary.
* Pregnant or breastfeeding women. Females of childbearing potential must have a negative serum pregnancy test at screening and agree to use a double-barrier method of contraception throughout the study period.
* Have a cardiac pacemaker or other indwelling foreign object that are contraindicated for MR imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with microdose (<2.5 millicurie; mCi) 18F-Raltegravir-related adverse events as measured by clinical observation during single intravenous dose administration and PET/MR imaging | One imaging session within 1 to 6 hours following administration of 18F-Raltegravir
Whole-body distribution (coronal through pelvis) of radiolabeled 18F-Raltegravir as determined by PET-MR scanning and quantification of radiographic regions of interest (ROI) immediately following and up to 4 hours after drug administration. | One imaging session within 1 to 6 hours following administration of 18F-Raltegravir

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Henrich, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States